CLINICAL TRIAL: NCT05563207
Title: Shijiazhuang Pingan Hospital
Brief Title: Application of Health Education Path of Traditional Chinese Medicine Nursin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shijiazhuang Pingan Hospital (Other)
Responsible Party: Principal Investigator, Jianhua Zhang, Director, Shijiazhuang Pingan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ShijiazhuangPinganH
Record Dates: First submitted 2022-09-26; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; health education; traditional Chinese medicine nursing
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Health Education

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): Both groups of patients were given routine treatment, and were intervened by the same batch of nursing staff. Among them, patients in the control group were given intervention for TCM health education standard path. During chemotherapy, the patient's condition was closely observed, patiently listened to the patient's chief complaint, answered their questions, and instructed the patient to follow the doctor's instructions to prevent complications such as infection and bleeding.
  Interventions: Other: traditional Chinese medicine health education standard path
- observation group (Active Comparator): The patients in the observation group were given TCM health education standard path intervention. The contents of the health intervention mainly included: ① Graphic and text education;②Language education;③ Psychological education; ④Dietary education; ⑤ Complication education
  Interventions: Other: traditional Chinese medicine health education standard path; Other: The contents of the health intervention mainly included:Graphic and text education; Other: The contents of the health intervention mainly included:Language education; Other: The contents of the health intervention mainly included:Psychological education; Other: The contents of the health intervention mainly included:Dietary education; Other: The contents of the health intervention mainly included:Complication education

INTERVENTIONS:
Other: traditional Chinese medicine health education standard path — Both groups of patients were given routine treatment, and were intervened by the same batch of nursing staff.During chemotherapy, the patient's condition was closely observed, patiently listened to the patient's chief complaint, answered their questions, and instructed the patient to follow the doctor's instructions to prevent complications such as infection and bleeding.
Other: The contents of the health intervention mainly included:Graphic and text education — When the patient was admitted to the hospital, the responsible nurse had a comprehensive understanding of the patient's disease cognition and psychological state, and based on this, an individualized intervention plan was formulated. With the help of publicity boards, brochures and other forms of pictures and texts, to popularize the knowledge and precautions of disease treatment for patients
  Arms: observation group
Other: The contents of the health intervention mainly included:Language education — adopt one-to-one method to inform patients of the principles, effects and precautions of chemotherapy, eliminate patients' misunderstandings, and repeat language education for many times during the treatment process to strengthen patients' memory
  Arms: observation group
Other: The contents of the health intervention mainly included:Psychological education — guide patients to express their own emotions, according to the patient's personality, cultural background, etc., after communicating with family members and negotiating, selectively inform the patient's actual condition
  Arms: observation group
Other: The contents of the health intervention mainly included:Dietary education — instruct patients to follow the principles of light, easy to digest and balanced nutrition
  Arms: observation group
Other: The contents of the health intervention mainly included:Complication education — Actively inform patients about complications in advance, and guide their prevention methods, such as increasing water intake, avoiding activities of affected limbs after chemotherapy, etc. Patients with vomiting, hair loss and other adverse reactions are prone to negative emotions such as anxiety and depression , timely take corresponding measures and appease the patient, inform them that it is a normal phenomenon, and guide them to maintain a good attitude.
  Arms: observation group

SUMMARY:
To explore the effect of traditional Chinese medicine (TCM) health education standard path on the treatment of patients with acute myeloid leukemia (AML). A total of 60 patients with acute myeloid leukemia in Shijiazhuang Ping An Hospital were selected and divided into control group (n=30) and observation group (n=30) according to the time of admission. Both groups received the same chemotherapy, the control group received routine nursing, and the observation group received TCM health education standard path intervention. The scores of Self-rating Anxiety Scale (SAS), Self-rating Depression Scale (SDS), Spitzer Quality of Life Index (QLI), awareness of TCM health education standard path content and nursing satisfaction were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the hospital for the first time during the observation period
* patients who met the diagnostic criteria for AML
* patients with stable disease, clear consciousness, fluent speech, and normal communication
* patients who volunteered to participate in the research

Exclusion Criteria:

* patients who were repeatedly admitted to hospital during the investigation period
* patients with hospitalization time ≤3 days
* patients whose condition changed after admission and could not continue to cooperate with the investigation
* patients who asked to withdraw during the observation period.

Ages: 37 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Self-rating anxiety scale | 3 months of intervention
  evaluate the anxiety of the two groups of patients before and after intervention
self-rating depression scale | 3 months of intervention
  evaluate depression of the two groups of patients before and after intervention
Quality of Life Index | 3 months of intervention
  the Spitzer Quality of Life Index (QLI) was used to evaluate the quality of life of patients
Self-made questionnaires to compare the awareness of traditional Chinese medicine health education standard path content | 3 months of intervention
  5 items of propaganda and education content, propaganda and education form, professional level of propaganda and education, nurses' professional attitude, and propaganda and education effect
Self-made questionnaires to compare nursing satisfaction | 3 months of intervention
  evaluate the nursing attitude, nursing skills, and explanations of medical staff

CONTACTS AND LOCATIONS:
Locations (1):
- Shijiazhuang Pingan Hospital, Shijiazhuang, Hebei, China